CLINICAL TRIAL: NCT00301769
Title: A Phase I Study of SJG-136 in Patients With Advanced Leukemia
Brief Title: SJG-136 in Treating Patients With Relapsed or Refractory Acute Leukemia, Myelodysplastic Syndromes, Blastic Phase Chronic Myelogenous Leukemia, or Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00100; NCI-2009-00100 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000462379; 2005-0607 (Other: M D Anderson Cancer Center); 6934 (Other: CTEP); U01CA062461 (NIH)
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Blastic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Chronic Lymphocytic Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Congenital Abnormalities; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — 1,1'-((propane-1,3-diyl)dioxy)bis(7-methoxy-2-methylidene-1,2,3,10,11,11a-hexahydro-5H-pyrrolo(2,1-c)(1,4)benzodiazepin-5,11-dione)

ARMS (1):
- Arm I (Experimental): Patients receive SJG-136 IV over 15 minutes on days 1-5. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of SJG-136 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A total of 10 patients are treated at the MTD.
  Interventions: Drug: SJG-136

INTERVENTIONS:
Drug: SJG-136 — Given IV

SUMMARY:
This phase I trial is studying the side effects and best dose of SJG-136 in treating patients with relapsed or refractory acute leukemia, myelodysplastic syndromes, blastic phase chronic myelogenous leukemia, or chronic lymphocytic leukemia. Drugs used in chemotherapy, such as SJG-136, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Establish the maximum tolerated dose of SJG-136 in patients with relapsed or refractory acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL) myelodysplastic syndrome (MDS), chronic myelogenous leukemia in blastic phase (CML-BP), or chronic lymphocytic leukemia (CLL).

II. Determine dose-limiting toxicities and pharmacokinetics of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive SJG-136 IV over 15 minutes on days 1-5. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of SJG-136 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A total of 10 patients are treated at the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following hematologic malignancies:

  * Acute myeloid leukemia
  * Acute lymphoblastic leukemia
  * Myelodysplastic syndromes
  * Chronic myelogenous leukemia in blastic phase
  * Chronic lymphocytic leukemia
* Relapsed or refractory disease
* No immediately available, potentially curable options (e.g., stem cell transplantation) available
* Bilirubin normal (unless elevated due to Gilbert's syndrome)
* HIV positivity allowed provided CD4 counts are normal with no AIDS-defining disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit study compliance
* Recovered from prior therapy
* ECOG performance status =< 2
* SGOT and SGPT =< 2.5 times upper limit of normal (ULN)
* Creatinine normal OR creatinine clearance >= 60 mL/min
* Primary resistance (i.e., failed to achieve a complete remission [CR] to a standard induction regimen) or relapsed after achievement of a CR.
* Must have documented failure to last cytotoxic regimen prior to study entry.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* No known CNS disease
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to SJG-136
* More than 7 days since radiotherapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other anti-leukemia agents except hydroxyurea =< 5 grams/day =< 14 days prior to and during first course of treatment to control blood counts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-12; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) determined according to dose-limiting toxicities (DLTs) graded using Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States